CLINICAL TRIAL: NCT02836119
Title: Sleep Behaviour and Gut Microbiota in Healthy Infants
Brief Title: Infant Sleep Behaviour and Gut Microbacteria
Acronym: SDEGU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Collaborators: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-00730
Record Dates: First submitted 2016-07-11; First posted 2016-07-18 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Gut Microbiota and Sleep in Infants
Keywords: Gut Microbiota; Gut Microbiome; Sleep; Infancy; Development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Stool samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The overarching study aim is to evaluate the development of sleep behavior and gut microbiota (GMB), and their potential interaction, during the vulnerable period of the first year of life. Age-specific fecal profiles with bacterial genome sequencing will provide new insight into the functional coevolution of the GMB and host sleep behavior.

ELIGIBILITY:
Inclusion Criteria:

* Good general health status
* exclusively breastfed (at baseline)
* vaginal birth delivery mode

Exclusion Criteria:

* C-section delivery mode
* Formula fed (at baseline)
* Diseases or lesions of the central nervous system, acute pediatric disease, developmental/neurologic/metabolic disorders, chronic medical conditions, or head injury
* Family history of narcolepsy/psychosis/bipolar disorder
* Conceptual age of < 37 or > 42 weeks
* Low birth weight (< 2500g)
* Co-sleeping during > 50% of the time in the same bed
* Medication use affecting sleep/alertness
* Vaccination (2 weeks prior to study)
* Antibiotics (3 months prior to study)
* Travelling across a time zone (within 1 month prior to study)
* intrauterine drug exposure, intrauterine infection, known or suspected drug or alcohol abuse
* Insufficient knowledge of German (parents)

Ages: 2 Months to 13 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy infants
Sampling Method: Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2016-07; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Differences in sleep phenotypes (high fragmentation vs low fragmentation, short vs long sleepers) | across the first twelve months of life
Differences in Gut Microbiome Diversity (alpha, beta, Shannon) and taxa abundance and association with sleep phenotypes | across the first twelve months of life

SECONDARY OUTCOMES:
Association of primary outcome measures with cognitive and behavioral questionnaires (Food, development, Sleep) | across the first twelve months of life

CONTACTS AND LOCATIONS:
Overall Officials: Salome Kurth, Dr. sc. nat., Principal Investigator — Clinic for Pulmonology
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No